CLINICAL TRIAL: NCT03208257
Title: Esmolol to Control Adrenergic Storm in Septic Shock- ROLL-IN 2
Acronym: ECASSS-R2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samuel Brown (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor-Investigator, Samuel Brown, Associate Professor, Pulmonary and Critical Care Medicine, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1050522
Record Dates: First submitted 2017-07-02; First posted 2017-07-05 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Septic Shock
Keywords: esmolol; adrenergic storm; septic shock
MeSH Terms: conditions — Shock, Septic | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Esmolol (Experimental): Intravenous esmolol will be administered as a continuous infusion according to protocol to control tachycardia with maximal infusion rates in the range of 10-40 mcg/kg/min.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — Esmolol hydrochloride infusion
  Other Names: BREVIBLOC

SUMMARY:
Septic shock is a common syndrome caused by the body's response to an infection. Septic shock is responsible for 10% of all ICU admissions and 30% of ICU deaths. Use of "beta blocker" medications may improve outcomes after septic shock. This pilot study evaluates protocols to infuse the beta blocker esmolol in patients with septic shock.

DETAILED DESCRIPTION:
This is a prospective, single arm, feasibility study of esmolol infusion in septic shock. The objective is to evaluate the feasibility, adequacy, and efficiency of study protocols for a subsequent ECASSS study. This study (ECASSS-R2) extends observations made in an initial pilot, ECASSS-R.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Within 72 hours of admission to the ICU and septic shock (sepsis present at time of admission)

   a. Septic shock defined by SEPSIS-3 consensus criteria as i. Suspected or documented infection ii. Sequential Organ Failure Assessment (SOFA) score increased by at least 2 points over baseline iii. Lactate > 2mmol/L iv. Receiving vasopressors to treat hypotension after at least 20 ml/kg intravenous crystalloid volume expansion
3. Receiving vasopressors through a central venous catheter for more than 60 minutes.
4. Arterial catheter in place or expected to be placed imminently.
5. Heart rate > 90/min while receiving vasopressors for more than 60 minutes.
6. Adequately volume expanded, as manifest by any of the following, performed as part of routine clinical care (i.e., no study procedures will be performed before signed consent). If none of these measures are clinically available, the clinical attending must confirm that volume expansion is adequate. (After enrollment, a final safety check will confirm the adequacy of volume expansion.)

   1. Central venous pressure (CVP) > 15 mm Hg.
   2. Negative Passive-Leg Raise (PLR) maneuver (<10% increase in cardiac output after PLR).
   3. No cardiac output response (<10% increase) after rapid infusion (<5 min) of 250 ml of IV crystalloid (i.e., a graded volume expansion challenge [GVEC]).
   4. Inferior vena cava (IVC) plethora
   5. For patients who happen to be breathing passively (i.e., paralyzed or deeply sedated) on a positive pressure mechanical ventilator delivering at least 8 ml/kg tidal volumes and in normal sinus rhythm, stroke volume variability <13% (such patients are acknowledged to be uncommon; the protocol does not recommend or require the induction of passive breathing).

Exclusion Criteria:

1. Lack of informed consent.
2. Currently receiving ExtraCorporeal Membrane Oxygenation (ECMO).
3. Known pregnancy or nursing.
4. Patient is a prisoner.
5. Patient on hospice (or equivalent comfort care approach) at or before the time of enrollment.
6. Known or current atrial fibrillation.
7. Previously enrolled in the trial.
8. Known allergy to esmolol or vehicle (see Appendix 2 for BREVIBLOC vehicle ingredients).
9. Receipt of nodal blocking agents (see Appendix 3 for list of such agents) within three half lives
10. Hemoglobin < 7 gm/dl.
11. Cardiac arrest within 24 hours.
12. Pulmonary hypertension (moderate or severe), from documented history of prior right heart catheterization or current evidence on transthoracic echocardiogram (TTE) of any of the following

    * Mean Pulmonary Arterial Pressure (mPAP) ≥ 35mmHg (millimeters of mercury)
    * Systolic Pulmonary Arterial Pressure (SPAP) ≥ 60mmHg (millimeters of mercury)
13. Cardiovascular collapse, as manifested by inability to achieve a mean arterial pressure (MAP) of 65 mmHg with vasopressor therapy.
14. Cardiogenic shock, as defined by any of the following

    * Cardiac index ≤ 2.3 L/min/m2
    * Ejection fraction ≤ 30%
    * ScvO2 ≤ 60%
    * Current infusion of any dose of dobutamine, milrinone, or dopamine (if dopamine is being used for clinically diagnosed bradycardia or cardiogenic shock)
    * Current infusion of epinephrine for clinically diagnosed cardiogenic shock
15. Significant atrioventricular dysfunction

    * Sick sinus syndrome
    * PR interval > 200 msec
    * Current evidence or prior history of Grade 2 or Grade 3 heart block
    * Pacemaker or plans to place a pacemaker
16. Pheochromocytoma or status asthmaticus
17. Receiving clonidine, guanfacine, or moxonidine
18. Worse than moderate aortic stenosis

    * Known aortic stenosis, with any of (1) mean gradient ≥ 40 mmHg OR (2) maximum gradient ≥ 60mmHg OR (3) aortic valve area ≤ 1.0cm2 OR (4) aortic valve area index ≤ 0.85cm2/m2 body surface area.
19. Worse than mild mitral stenosis

    * Known mitral stenosis, with any of (1) valve area ≤ 1.5 cm2 OR mean gradient ≥ 5 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Organ-failure-free days | 28 days

SECONDARY OUTCOMES:
All-cause hospital mortality | During hospitalization
All-cause 28-day and 90-day mortality | 28 days and 90 days
Peak serum high-sensitivity troponin | 24 hours
Left ventricular (LV) longitudinal strain | 24 hours
ICU-free days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M Brown, MD MS, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
In order to protect patient privacy and comply with relevant regulations, identified data will be unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code